CLINICAL TRIAL: NCT02408094
Title: Screening Sensitive Protein Markers and Exploring Application in Syndrome Diagnosis of Hot-dampness and Blood Stasis Syndrome in Patients With Rheumatoid Arthritis
Brief Title: Screening Protein Markers in Patients With Rheumatoid Arthritis and Hot-dampness and Blood Stasis Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Juan Jiao, Attending physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 81403364
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Heat-dampness and blood stasis syndrome; Protein markers
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to explore the protein markers and to applicate those protein markers in syndrome diagnosis of hot-dampness and blood stasis syndrome in patients with RA.

DETAILED DESCRIPTION:
RA is one of the main disabling diseases in nowadays, which is an autoimmune disease with complex networks mechanism involving multiple signaling pathways and existing cross path. The investigators consider that the "heat-dampness and blood stasis" syndrome is the main syndrome and major pathogenesis for active RA, which on the base of the theory of traditional Chinese medicine and a large quantity of clinical practice, and also examined by mechanism experiments. But the material basis of this syndrome is remained unclear, lack of high specific objective basis to ensure the syndrome differentiation consistency accurately in clinical practice. Proteomic techniques study cells or the body by all the protein expression and function, thus has the potential efficient for decoding syndrome biological basis. Proteomic techniques are the most effective way to reveal the essence of TCM syndrome. The investigators will use proteomic technology to explore the protein markers and to applicate those protein markers in syndrome diagnosis of hot-dampness and blood stasis syndrome in patients with RA. With strong clinical applicability, this will reveal the scientific connotation of this syndrome, preliminarily guide the syndrome differentiation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are made or confirmed diagnosis according to the American College of Rheumatology criterion and "heat-dampness and blood stasis" syndrome according to Traditional Chinese Medicine.

Exclusion Criteria:

1. Subjects have other serious diseases, such as liver and kidney disease, cerebral-cardio vascular diseases.
2. Subjects, who belong to "non-heat-dampness and blood stasis" syndrome, have double syndrome of heat or dampness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with rheunmtoid arthritis and "heat-dampness and blood stasis" syndrome
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
serum and saliva protein markers | six hours

CONTACTS AND LOCATIONS:
Overall Officials: Jiao Juan, Doctor, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided